CLINICAL TRIAL: NCT02369692
Title: Embolization Procedures in the Peripheral Vasculature Using the Magellan™ Robotic System
Status: Terminated | Type: Observational
Sponsor: Hansen Medical (Industry)
Responsible Party: Sponsor
Other Study IDs: HMP 021 Embolization
Record Dates: First submitted 2015-02-06; First posted 2015-02-24 (Estimated); Last update posted 2018-03-01 (Actual); Status verified 2015-09

CONDITIONS: Peripheral Vascular Disease
MeSH Terms: conditions — Peripheral Vascular Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Magellan Robotic 6 Fr Catheter — The Hansen Medical Magellan™ Robotic Catheter 6 Fr (Magellan™)

SUMMARY:
The purpose of this prospective study is to gather procedural use and safety data on the initial use of the Magellan Robotic System with the Magellan Robotic Catheter 6 Fr, Vascular Accessories 6 Fr and Microcatheter Driver This study will focus on, but not be limited to, endovascular embolization procedures in the peripheral vascular, for example, embolization of the splenic and hepatic arteries, uterine arterial embolization (UAE), prostatic arterial embolization (PAE), and trans-arterial chemoembolization (TACE).

The data will be analyzed for medical education, societal presentation and/or publication by the investigator.

DETAILED DESCRIPTION:
The primary objectives of this study are to evaluate the safety and clinical performance of the Magellan Robotic System with the 6 Fr catheter, Vascular Accessories 6 Fr and Microcatheter Driver in patients who are indicated for an embolization procedure or other endovascular procedure in the peripheral vasculature.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Able and willing to provide written informed consent
* Eligible for an embolization procedure or other endovascular procedure in the peripheral vasculature
* Not participating in an investigational study involving the peripheral vasculature

Exclusion Criteria:

* Vasculature cannot accommodate the Magellan Robotic Catheter or required accessories
* The required delivery of therapeutic device(s) "through" the Magellan Robotic Catheter in which the diameter for the therapeutic device(s) is/are incompatible with the Magellan Robotic Catheter
* An endovascular approach to the treatment of peripheral vasculature disease is contraindicated
* Sepsis
* Major coagulation abnormalities
* Presence of significant co-morbid illness that contraindicates surgery or an interventional radiological procedure
* Unmanageable contrast agent hypersensitivity
* Patients who are prisoners
* Patients who are mentally incapacitated, e.g., comatose, unresponsive, cannot provide informed consent, or are deemed unreliable or unstable by the investigator or with a cognitive impairment
* Pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A subject must be a candidate for an embolization procedure or other endovascular procedure in the peripheral vasculature, meet all inclusion and no exclusion criteria, and be willing to comply with all protocol testing and follow-up.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2014-04; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Evaluation of Safety and Clinical Performance of the Magellan Robotic system with the 6 Fr Catheter. (incidence and description of reported Magellan System device related or contributed adverse events and device deficiencies) | 2 Days
  The primary performance endpoint is device success defined as successful cannulation of the target blood vessel with the Magellan Robotic Catheter 6 Fr, Vascular Accessories 6 Fr and Microcatheter Driver on the first attempt, then accurate delivery of therapy.
  The primary safety endpoint is the incidence and description of reported Magellan System device related or contributed adverse events and device deficiencies through the study period.
Device success (Successful cannulation of the target blood vessel with the Magellan Robotic Catheter 6 Fr, Vascular Accessories 6 Fr and Microcatheter Driver on the first attempt, the accurate delivery of Therapy) | 2 Days
  Successful cannulation of the target blood vessel with the Magellan Robotic Catheter 6 Fr, Vascular Accessories 6 Fr and Microcatheter Driver on the first attempt, the accurate delivery of Therapy

SECONDARY OUTCOMES:
Number of Participation with Adverse Events | 30 days
  To evaluate use of the leader of Microcatheter as primary device for deliver of the therapy

CONTACTS AND LOCATIONS:
Overall Officials: Brenda Cayme, RN, BSN, Study Director — Hansen Medical Inc
Locations (1):
- Hôpital Européen Georges Pompidou, Paris, France